CLINICAL TRIAL: NCT04064463
Title: Dual Reinforcement Contingency Management for Alcohol Use Disorders
Acronym: Peth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sheila Alessi, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-146-2
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder; Contingency Management
MeSH Terms: conditions — Alcoholism | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Standard care
  Interventions: Behavioral: Standard care
- Experimental Group (Experimental): Standard care plus contingency management
  Interventions: Behavioral: Standard care; Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Standard care — standard treatment for substance use disorders, along with sample monitoring
Behavioral: Contingency management — Participants can earn reinforcement for attending group and abstinence from alcohol
  Arms: Experimental Group

SUMMARY:
Phosphatidylethanol (PEth) is a direct biomarker of alcohol that can detect moderate to heavy drinking with high sensitivity and specificity over 3-week periods. Reinforcing negative PEth results alongside attendance may increase the proportion of participants who respond to CM during and post treatment. In the proposed study, the investigators will collect PEth samples every 3 weeks for 12 weeks in 150 participants initiating outpatient treatment for alcohol use disorders. Using a two-group randomized design, participants will be assigned to standard care with PEth monitoring alone or with CM for attending treatment and submitting PEth negative samples. Compared to standard care and monitoring, the investigators expect that the CM intervention will result in greater attendance, more PEth negative samples, and higher proportions of self-reported non-drinking days, along with lower proportions of heavy drinking days, over the short term and the long term, measured throughout a 12-month follow-up. The investigators anticipate that the reinforcement intervention may decrease other drug use and sexual risk behaviors that spread HIV, reduce psychiatric symptoms, and improve quality of life as well.

ELIGIBILITY:
Inclusion Criteria:

* in intensive outpatient treatment
* DSM-5 diagnosis of an alcohol use disorder

Exclusion Criteria:

* have a condition that may hinder study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Group attendance | 12 weeks
  longest consecutive days attended groups
Alcohol abstinence | 12 weeks
  number of negative PEth samples

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Alessi, Ph.D., Principal Investigator — UConn Health
Locations (1):
- The Village, Hartford, Connecticut, United States